CLINICAL TRIAL: NCT01671930
Title: Maastricht Biomarker CT Study. Relation Between Cardiovascular Biomarkers and Coronary Atherosclerosis in Patients Undergoing Multi Detector Cardiac Computed Tomography.
Brief Title: Maastricht Biomarker CT Study
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MEC 08-4-057
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Artery Disease; Coronary Stenosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiac computed tomographic angiography: Patients refered for cardiac computed tomographic angiography by a cardiologist.

SUMMARY:
Introduction

Cardiovascular disease is the leading cause of death in the Western world. The main cause for cardiovascular events is the development of atherosclerosis in the coronary arteries. In more than 70% of cases, myocardial infarctions are caused by atherosclerotic plaque rupture, which results in subsequent formation of an occluding thrombus. Plaques that have a high risk of rupture are called vulnerable plaques. Cardiovascular imaging provides a complementary diagnostic approach in the assessment of cardiovascular risk in patients. However, the lack of biological detection possibilities of current imaging technologies limits their predictive value. For instance, multi detector computed tomography (MDCT) is an excellent tool to visualize coronary atherosclerosis. However, individual risk assessment is still problematic. Which of the diagnosed atherosclerotic plaques will undergo plaque rupture and lead to acute vascular events is currently hard to predict. Potentially, serum biomarkers could help identify the patient at risk. A wide variety of prognostic markers related to atherosclerosis have been identified in the past to predict for cardiovascular events. Nevertheless, their predictive value in individual patients is still limited. A difficulty in serum biomarker research is the requirement of large patient cohorts to study the relation between event rate and serum biomarker levels. The necessity to perform lengthy and costly studies, hinders the translation of novel cardiovascular serum biomarkers into the clinic. An alternative approach could be to study the correlation between levels of serum biomarkers and the presence of atherosclerosis in the coronary arteries.

Study objectives

Primary objective of the present analysis is to investigate the predictive value of a variety of serum biomarkers to predict atherosclerosis in the coronary tree of patients undergoing cardiac MDCT.

Design and Methods

Patients undergoing cardiac MDCT are eligible for the study. Excluded are patients with acute coronary syndrome, hemodynamic instability, pregnancy, severe renal insufficiency, allergy for contrast medium and inability to obtain informed consent. Permission to store the serum samples for future analysis of new prognostic markers for cardiovascular events will be acquired from the patients. Written information is send to the patient at least 1 week prior to CT. The samples will be stored coded, at the Biobank Maastricht, for a maximum duration of 15 years. Once measurements from the samples will be performed, the serum samples will be sent by the Biobank coded to the analyzing researchers, which have no access to the key file where codes are linked to the specific hospital identity number. This file will be stored by an independent researcher at the Cardiology department of the Maastricht University Medical Center. The assessment of atherosclerotic burden of the coronary tree will be performed by cardiac MDCT specialists blinded to the clinical data and serum biomarker outcome. Biomarker levels are correlated to the severity and amount of coronary artery disease as assessed by cardiac MDCT.

ELIGIBILITY:
Inclusion Criteria:

* patients refered to cardiac computed tomography to exclude coronary artery disease

Exclusion Criteria:

* pregnancy
* severe renal insufficiency
* severe allergy to contrast medium
* Inability to obtain informed consent
* Age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that were refered to undergo cardiac computed tomography by their cardiologist, to exclude coronary artery disease. Location: tertiary academic hospital.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2007-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
coronary artery disease | 1 year
  * The presence of any coronary atherosclerotic plaque as visible on cardiac CT.
  * The presence of any significant (≥50% luminal stenosis) coronary plaque in the coronary tree.
  * The number of atherosclerotic plaques in the coronary tree.
  * The calcium score (Agatston method).
  * Plaques are categorized as calcified (exclusively content with density >130 Hounsfield units), non-calcified (exclusively content with density <130 Hounsfield units), or mixed (characteristics of both calcified and non-calcified plaque).

CONTACTS AND LOCATIONS:
Overall Officials: H Crijns, M.D. P.h.D., Principal Investigator — Maastricht University Medical Center; B Kietselaer, M.D. P.h.D., Study Director — Maastricht University Medical Center; L Hofstra, M.D. P.h.D, Study Chair — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Background] Mingels AM, Joosen IA, Versteylen MO, Laufer EM, Winkens MH, Wildberger JE, Van Dieijen-Visser MP, Hofstra L. High-sensitivity cardiac troponin T: risk stratification tool in patients with symptoms of chest discomfort. PLoS One. 2012;7(4):e35059. doi: 10.1371/journal.pone.0035059. Epub 2012 Apr 25. PMID 22558116
- [Result] Laufer EM, Mingels AM, Winkens MH, Joosen IA, Schellings MW, Leiner T, Wildberger JE, Narula J, Van Dieijen-Visser MP, Hofstra L. The extent of coronary atherosclerosis is associated with increasing circulating levels of high sensitive cardiac troponin T. Arterioscler Thromb Vasc Biol. 2010 Jun;30(6):1269-75. doi: 10.1161/ATVBAHA.109.200394. Epub 2010 Mar 18. PMID 20299689
- [Derived] de Wit-Verheggen VHW, Altintas S, Spee RJM, Mihl C, van Kuijk SMJ, Wildberger JE, Schrauwen-Hinderling VB, Kietselaer BLJH, van de Weijer T. Pericardial fat and its influence on cardiac diastolic function. Cardiovasc Diabetol. 2020 Aug 17;19(1):129. doi: 10.1186/s12933-020-01097-2. PMID 32807203